CLINICAL TRIAL: NCT00302822
Title: Enfuvirtide for the Initial Phase of Antiretroviral Therapy in HIV-infected Patients With High Risk of Clinical Progression : ANRS 130 APOLLO
Brief Title: Intensification With Enfuvirtide in Naive HIV-infected Patients (ANRS130)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Collaborators: Hoffmann-La Roche (Industry); Gilead Sciences (Industry)
Responsible Party: Sponsor
Organization: ANRS, Emerging Infectious Diseases (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005-004722-12; 2005-004722-12 (EudraCT Number)
Record Dates: First submitted 2006-03-14; First posted 2006-03-15 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2013-07

CONDITIONS: HIV Infections; AIDS
Keywords: HIV infections; Fuzeon; Truvada; AIDS; Treatment Naive
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Enfuvirtide; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Lopinavir; efavirenz; lopinavir-ritonavir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intensification (Experimental): lopinavir or efavirenz and emtricitabine/tenofovir and intensification with enfuvirtide (week 0 to 24)
  Interventions: Drug: enfuvirtide; Drug: emtricitabine/tenofovir; Drug: lopinavir or efavirenz
- Standard (Active Comparator): lopinavir or efavirenz and emtricitabine/tenofovir
  Interventions: Drug: emtricitabine/tenofovir; Drug: lopinavir or efavirenz

INTERVENTIONS:
Drug: enfuvirtide — from week 0 to 24
  Other Names: Fuzeon
  Arms: Intensification
Drug: emtricitabine/tenofovir — 1 pill/day
  Other Names: Truvada
Drug: lopinavir or efavirenz — investigator choice
  Other Names: Kaletra, Sustiva

SUMMARY:
HIV infection is diagnosed late in a substantial proportion of patients having an increased risk of clinical progression (AIDS, new AIDS-defining event or death). The currently recommended antiretroviral therapy has suboptimal activity in this setting and potent quadruple-drug therapy has not been sufficiently evaluated. Enfuvirtide may be an appropriate candidate as the fourth antiretroviral agent, regarding its activity, its parenteral administration avoiding gastrointestinal symptoms that often lead to interruption of treatment, the lack of pharmacokinetic interactions and the absence of systemic toxicity.

The aim of this study is to investigate, in a comparative intensification trial, the immunological benefit of adding enfuvirtide for 6 months to a conventional antiretroviral therapy in HIV-1 infected and severely immunosuppressed patients, naïve of any antiretroviral treatment.

We postulate that addition of enfuvirtide to a first-line antiretroviral therapy consisting in emtricitabine/tenofovir combined with either efavirenz or lopinavir/r may improve immunological restoration, measured as the proportion of patients with more than 200 CD4 cells per mm3 after 24 weeks of antiretroviral therapy.

DETAILED DESCRIPTION:
The purpose of this randomized, open-label study is to evaluate the immunological efficacy of two first-line strategies of antiretroviral therapy:

1. emtricitabine/tenofovir disoproxil fumarate coformulated plus efavirenz (or lopinavir/r) intensified by enfuvirtide during the first 24 weeks of therapy.
2. emtricitabine/tenofovir disoproxil fumarate coformulated plus efavirenz (or lopinavir/r)

Patients with lymphocytes T CD4+ cell (CD4)count below 100 per mm3, or CD4 cell count below 200 per mm3 and past history or presence of AIDS defining event and naïve of any antiretroviral therapy will be eligible. This multicenter study will enroll 220 patients (n=110 in each arm). The planned duration of the study is 48 weeks from the enrolment of the last subject.

The primary endpoint will be immunological success defined as CD4 cell count above 200 cells per mm3 after 24 weeks of initial treatment. The durability of this response will be evaluated and patients will be followed for 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Antiretroviral naïve HIV-1 infected patients
* CD4 cell count below 100 per mm3, or CD4 cell count below 200/mm3 and past history or presence of B or C(AIDS defining)event
* Signed informed consent

Exclusion Criteria:

* Pregnancy; breast feeding
* Coinfection with HIV-2 or infection with HIV-1 subtype O
* Antiretroviral pretreated patients
* Neoplasia disease currently treated with chemotherapy or radiotherapy
* Severe liver failure
* Treatment with cytokines or HIV vaccine trial
* One or more of the following biological abnormalities: hemoglobin below 10 g/dl, Neutrophils below 750 per mm3, thrombocytopenia below 50000 per mm3, creatinine clearance below 60 ml per min, Liver Function Tests over 3 Upper Limit of Normal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2006-04; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Immunological success defined as a CD4 cell count above 200 cells per mm3 after 24 weeks of initial antiretroviral treatment | 24 weeks

SECONDARY OUTCOMES:
Virological response, clinical progression, tolerance,toxicity, quality of life under therapy, adherence and resistance mutations emerging in case of virological failure. | from 0 to 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Veronique Joly, MD, Principal Investigator — Hopital Bichat Claude Bernard Paris France; Geneviève Chêne, MD PHD, Study Director — INSERM U897 Bordeaux France
Locations (1):
- Service des Maladies Infectieuses A Hôpital Bichat-Claude Bernard, Paris, France